CLINICAL TRIAL: NCT04910633
Title: Medical Treatment of Solid Tumors at the Lyon University Hospital Cancer Institute During the First Wave of COVID-19 in France: A Conservative Approach
Acronym: COCA
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_0005
Record Dates: First submitted 2021-05-10; First posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Cancer; Solid Tumor; Covid19
Keywords: COVID-19; Cancer; Solid Tumor; Qualitative study; First pandemic wave
MeSH Terms: conditions — Neoplasms; COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Solid Tumor and COVID-19: Patients with a solid tumor followed by an oncologist of Lyon University Hospital Cancer Institute (LUHCI) who have been hospitalized at LUHCI for the COVID-19 between March and May 2020 and who didn't oppose the reuse of their medical file data for research purpose.
  Interventions: Other: COCA is an observational study based on retrospective data issued from patient medial file.

INTERVENTIONS:
Other: COCA is an observational study based on retrospective data issued from patient medial file. — The following parameters will be collected from the medical files of the patients involved in this study:
  * Age
  * Gender
  * Cancer type
  * Cancer Stage
  * Cancer Treatment
  * COVID-19 severity (based on chest X-Ray damage. Low ≤25%, Middle: between 25-50%, High above 50%)
  * Living Status
  * Attribution of Mortality to COVID status
  * Comorbidities

SUMMARY:
An article to present how cancer patients were taken in charge at Lyon University Hospital Cancer Institute (France) during the first peak of the COVID-19 pandemic between March and May 2020 is under writing.

It will present strategies that were set-up to avoid cross-contamination between patients and caregivers, patients treatment adaptation (timing, dosage,..) and how consultations, multidisciplinary team meetings, surgical procedures and clinical trials were impacted.

Part of this article will also illustrate the characteristics of patients with a solid tumor(s) that have been hospitalized during this timeframe for the COVID-19. How cancer type and stage affect Covid severity and mortality.will be described for a small sample of patients (44). These qualitative figures will be compared to literature current state of the art.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a LUHCI code created after 2015 and a LUHCI COVID-19 code created between March 2020 and May 2020.

Exclusion Criteria:

* Patients who did not allow the reuse of their medical file data for research related to COVID-19-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a LUHCI cancer code created after 2015 and a LUHCI COVID-19 code created between March 2020 and May 2020.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2021-01-22 (Actual)

PRIMARY OUTCOMES:
Illustration of the repartition of COVID+ patient severity (Low/Medium/Severe status) depending on cancer nature, stage and patient age. | At the end of Month 1
  COVID-19 severity will be determined based on chest X-Ray damage as follow. Low severity : ≤25% of chest X-Ray damage, Middle severity: between 25-50% of chest X-Ray damage, High Severity : above 50% of chest X-Ray damage.
  A graphic will then be drafted to present the relationship between Covid-19 severity depending on patient age, cancer nature, and cancer stage.

CONTACTS AND LOCATIONS:
Locations (1):
- Lyon University Hospital Cancer Institute, Bron, France